CLINICAL TRIAL: NCT06491992
Title: Effect of Chitosan Phonophresis on Cervical Pain and Disability in Smartphone Addicted Users
Brief Title: Chitosan Phonophresis on Cervical IN Smartphone Addicted Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lama Saad El-Din Mahmoud, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O6U.PT.REC/024/002003
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Chitosan Phonophresis intervention
  Interventions: Drug: Chitosan Phonophresis; Other: selected physical therapy exercise
- control group (Experimental): the selected exercise program
  Interventions: Other: selected physical therapy exercise

INTERVENTIONS:
Drug: Chitosan Phonophresis — Chitosan Phonophresis, three times per week for four weeks.
  Arms: study group
Other: selected physical therapy exercise — selected neck exercise and electrotherapy on cervical region

SUMMARY:
A phonophoresis-based drug delivery system is a synchronous approach to improve local drug penetration in neuromuscular diseases associated with neuronal damage, excruciating pain, and local inflammation. Chitosan, a semi-synthetic material, is obtained by partial deacetylation of chitin amines, resulting in copolymers of N-acetylglucosamine and N-glucosamine. Its use has been explored in various biomaterial and medical applications. Chitosan has emerged as a cost-effective, biocompatible, and biodegradable material with many desirable biological properties, improvement of homeostasis and antiviral potential. Chitosan was found to suppress pro-inflammatory cytokines and decreased peripheral nerve edema, the polycationic nature of chitosan allows it to absorb protons, which reduces inflammation and provides an analgesic effect.

DETAILED DESCRIPTION:
The patients will randomly be divided into two equal groups; the control group which will receive the selected exercise program and the study group will receive the same exercise training program in addition to Chitosan Phonophresis, three times per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranged from 16-18 years
* body mass index will be 26.58 kg/m2.
* used a smart phone for more than 1 year for at least 2 hours per day
* complaining of neck pain after using a smart phone, addiction to smart phone in accordance with the smart phone addiction scale (SAS)

Exclusion Criteria:

* any previous head and neck injuries or surgeries
* any congenital abnormalities or symptomatic deformity in either the cervical or the lumbar spine
* any uncorrected visual or auditory problems, dizziness, vertigo and headache
* any systematic diseases, any addiction to alcohol, any additive drugs and sedatives within 48 hours previous to tests
* body mass index of subjects over25 kg/m2.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Version (SAS-SV) | four weeks
  SAS-SV was psychometrically robust in measuring the severity of smartphone addiction
The visual analogue scale | four weeks
  was utilized to evaluate pre- and post-treatment neck pain
Neck disability index | four weeks
  assess how neck pain and other symptoms manifested during various functional activities. Ndi had been reported as a reliable (Cronbach's alpha: 0.89) and valid instrument to evaluate self-rated disability in patients with neck pain

SECONDARY OUTCOMES:
Cervical ROM | four weeks
  Cervical active ROM will be measured for each participant in the study by digital goniometer device.

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No